CLINICAL TRIAL: NCT01988857
Title: Safety and Reactogenicity of GSK Biologicals' dTpa Vaccine (Boostrix™) in Healthy Vietnamese Children
Brief Title: Safety of a Booster Dose of GlaxoSmithKline (GSK) Biologicals' Boostrix™ Vaccine in Healthy Vietnamese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 115739; 2013-003859-37 (EudraCT Number)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-06

CONDITIONS: Diphtheria; Tetanus; Acellular Pertussis
Keywords: Vietnam; Children; Reactogenicity; BoostrixTM; Safety; dTpa; Booster; Healthy
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Boostrix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dTpa Group (Experimental)
  Interventions: Biological: Boostrix™

INTERVENTIONS:
Biological: Boostrix™ — Single-dose administered intramuscularly in the deltoid region of non-dominant arm.

SUMMARY:
This study will evaluate the safety and reactogenicity of GSK Biologicals' combined reduced-antigen-content diphtheria-tetanus-acellular pertussis (dTpa) vaccine, Boostrix™ when given as a single injection to 6-10 year old children. Data that are available globally on the age group from four to six years of age will be used to bridge the age gap in this study and aid in the registration of the vaccine for children from the age of four years.

DETAILED DESCRIPTION:
A phase III, single-group, open-label study of GSK Biologicals' vaccine BoostrixTM administered as a booster vaccine dose in healthy Vietnamese children aged 6-10 years. A single booster dose of BoostrixTM will be administered at Visit 1 (Day 0) and subjects will be observed until Visit 2 (Day 30). Safety will be assessed in terms of solicited adverse events (during 4 days post vaccination), unsolicited adverse events (during 31 days post vaccination) and serious adverse event (during the trial period).

This protocol summary was updated following an administrative change of adding the EudraCT number to this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 10 years of age at the time of the vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Written informed assent to be obtained from the subject in addition to the informed consent signed by the parent(s)/LAR(s), as required by local regulations.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects who have previously completed their routine vaccinations against diphtheria, tetanus and pertussis diseases according to the local recommended vaccination schedule at that time and have not received the vaccine in the last two years prior to study dose administration.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced abstinence or adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to vaccination. Inhaled and topical steroids are allowed.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to the booster vaccine dose, or planned administration during the study period.
* Administration of immunoglobulins and/or any blood products within the three months preceding Visit 1 or planned administration during the study period.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* A history of previous or intercurrent diphtheria, tetanus or pertussis disease.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Major congenital defects or serious chronic illness.
* Acute disease and/or fever at the time of enrollment.
* Pregnant or lactating female.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2014-02-22 (Actual); Primary Completion 2014-05-10 (Actual); Study Completion 2014-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 302 subjects enrolled into the study, 2 were excluded due to developing allergic reactions and hence only 300 started the study.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Boostrix Group: Subjects received a single dose of Boostrix vaccine at 6-10 years of age.
Period: Overall Study
Arm/Group | Boostrix Group
Started | 300
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Boostrix Group
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 300
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.9 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian Heritage | 300

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. Relationship analysis was not performed.
Time Frame: Within 4 days (Days 0-3) post vaccination period
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group
Number analyzed (Participants) | 300
Participants
  Any Pain | 105
  Any Redness | 55
  Any Swelling | 40
  Grade 3 Pain | 1
  Grade 3 Redness | 1
  Grade 3 Swelling | 3

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache and temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 4 days (Days 0-3) post vaccination period
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group
Number analyzed (Participants) | 300
Participants
  Any Fatigue | 42
  Any Gastrointestinal symptoms | 15
  Any Headache | 33
  Any Temperature | 14
  Grade 3 Fatigue | 1
  Grade 3 Gastrointestinal symptoms | 0
  Grade 3 Headache | 0
  Grade 3 Temperature | 0
  Related Fatigue | 40
  Related Gastrointestinal symptoms | 14
  Related Headache | 33
  Related Temperature | 13

3. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 31 days (Days 0-30) post vaccination period
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group
Number analyzed (Participants) | 300
Participants | 19

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (From Day 0 to Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group
Number analyzed (Participants) | 300
Participants | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms during the 4-day (Days 0-3) post-vaccination period, Unsolicited AEs during the 31-day (Days 0-30) post-vaccination period, SAEs during the entire study period (from Day 0 to Day 30).
Arm/Group | Boostrix Group
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300
Other Adverse Events (participants affected / at risk) | 133/300
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Group (N=300)
Pain (General disorders) | 105
Redness (General disorders) | 55
Swelling (General disorders) | 40
Fatigue (General disorders) | 42
Gastrointestinal symptoms (General disorders) | 15
Headache (General disorders) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.